CLINICAL TRIAL: NCT04288271
Title: TAKE-IT TOO: Teen Adherence in KidnEy Transplant Improving Tracking To Optimize Outcomes
Brief Title: Teen Adherence in KidnEy Transplant Improving Tracking To Optimize Outcomes - Stage 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Bethany Foster, Chair of the Department of Pediatrics, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MP-CUSM-15-598; 5R01DK110737 (NIH)
Record Dates: First submitted 2017-12-18; First posted 2020-02-28 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Medication Adherence; Kidney Transplantation
Keywords: pediatric; adolescent; renal; allograft; immunosuppressive; immunosuppression; adherence; medication; young adult; mobile health; compliance; randomized trial; electronic pillbox
MeSH Terms: conditions — Medication Adherence; Patient Compliance

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants (patient-, parent- and HCP-participants) will be blinded to group allocation but, given the nature of the intervention, study coordinators who will be acting as coaches must be aware of group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adherence Intervention (Experimental): The objective of the intervention is to improve medication adherence. Patient-participants will use a multi-dose electronic pillbox and adherence tracking website which can provide dose reminders. Patient will form an Adherence Support Team (AST) including the participant, a parent (or other) and the "Coach" (study coordinator). The Coach will guide the AST to use Action-focused Problem-solving to address personal barriers to adherence. They will then generate concrete "if-then" plans for how they will behave in a given situation. Intervention participants with excellent adherence will be encouraged to work on building autonomy in medication-taking instead of adherence. Action plans will be able to be modified, if desired, at the 6-week and 10-week check-ins.
  HCP-participants at intervention sites will be given the option to login to the adherence tracking website to view the adherence data of their patients. They will also be alerted by study staff to critical non-adherence events.
  Interventions: Behavioral: Adherence Intervention
- Healthy Living Education Intervention (Other): Patient-participants will receive a healthy living education intervention with the use of an e-pillbox. Contacts with the coach will occur at the same intervals as at adherence intervention sites. Participants will choose one of 3 healthy living topics on which they will receive education in an interactive format. The coach will engage the participant in a semi-scripted conversation on the selected topic. At check-ins, the coach will either continue the conversation on the topic selected at the outset or provide education on another topic. The coach will NOT engage in discussions about adherence and will NOT provide feedback on adherence data.
  Interventions: Other: Healthy living education intervention

INTERVENTIONS:
Behavioral: Adherence Intervention — Intervention:
  * Adherence Support Team (patient, parent or a significant other, Coach)
  * Standardized educational videos on immunosuppressive medications, rejection, and improving adherence
  * Identification of adherence barriers, self-efficacy for medication-taking, and allocation of treatment responsibility
  * 'Action-Focused Problem-Solving' to address barriers selected as most important by the patient
  Device:
  * Electronic pillbox monitoring with text message and/or audio/visual dose reminders and access to e-pillbox website
  * Feedback of electronic monitoring data at increasing intervals between initiation of the intervention at 4-week and exit at 14-week.
  Other Names: Action-focused problem-solving; Electronic multi-dose pillbox monitoring system; Medy Box; Portable e-pillbox
  Arms: Adherence Intervention
Other: Healthy living education intervention — Intervention:
  * Standardized educational videos on immunosuppressive medications, rejection, and improving adherence
  * Healthy living topic discussion at increasing intervals between 4-wk and 14-wk visits
  * 'Action-Focused Problem-Solving' to address barriers on healthy living topic selected by the patient
  Device:
  • Electronic adherence monitoring without dose reminders or feedback (enrollment to 14w)
  Arms: Healthy Living Education Intervention

SUMMARY:
Medication non-adherence is a major problem in kidney transplant recipients; young people 12-24 years of age are at particularly high risk for non-adherence and graft failure compared to young children and adults. Given that poor medication contributes greatly to graft failure, clinically feasible and effective interventions are urgently needed to improve adherence, survival, and quality of life in this population. The broad aim of this prospective, 3-stage, sequential study is to improve medication adherence in adolescent kidney transplant recipients by: 1) adapting the successful Teen Adherence in Kidney transplant Effectiveness of Intervention Trial (TAKE-IT) intervention for use in 'real world' clinical care, 2) designing and testing a new portable electronic pillbox and companion tracking website interface, and 3) preliminary testing of the adapted intervention.

DETAILED DESCRIPTION:
This entry describes Stage 3 of the study. In Stage 3, the adapted intervention and new e-pillbox and adherence-tracking website will be piloted in preparation for a definitive cluster-randomized trial (CRT). This study builds on the lessons from TAKE-IT and is a critical step towards a scalable intervention for real-world use.

Stage 3 aims to pilot the adapted intervention, including the new e-pillbox, in a CRT to:

1. Determine the feasibility of a full-scale CRT (process considerations, attrition)
2. Understand all stakeholders' experience with the intervention, including the degree to which the e-pillbox and adherence-tracking website are integrated into daily life by patients and into practice by HCP
3. Estimate intra-cluster correlation coefficients (ICC) and other statistical parameters related to adherence outcomes relevant for sample size planning for a CRT. Adherence outcomes to be considered include daily proportion of patients with 100% taking adherence (defined as having taken all prescribed doses in a day) and daily proportion of patients with correct dosing (defined as having taken all prescribed doses within 2 hours before or after the scheduled time).

The adapted adherence-promoting intervention will be compared with another intervention in a pilot parallel-groups CRT. The interventions will be applied over 10 weeks. Participating centers, rather than patients, were randomized using a restricted randomization strategy with the Montreal Children's Hospital (MCH) assigned to the adherence intervention. This is necessary to ensure that the PI and lead site get sufficient experience with the intervention to guide other sites and to prepare for the full-scale CRT. All other sites were randomized, stratified on center size, to the new adherence intervention or the healthy living education intervention (control arm); this ensured adequate numbers of participants in each arm.

The aim is to enroll 67 patients across all sites over a 6-month interval. Based on numbers of available patients at each site, the targets noted above represent 13-50% of eligible patients at a given site. Allowing for 10% drop-out, 60 will complete the study (TAKE-IT had 4% drop-out by 6 mo.). Parents of eligible patients <18y old who have agreed to participate in the study will also be eligible to participate (57 parents anticipated). We will also enroll 2-3 HCPs, most involved with direct patient care, at each adherence intervention site to allow capture of information on their experience with the e-pillbox system and intervention over the course of the study (9 HCPs anticipated). No HCP will be enrolled at healthy living intervention sites. Participants will be blinded to group allocation but, given the nature of the intervention, coaches must be aware of group allocation.

Patients participants: Enrollment will be followed by a 4-week run-in period during which adherence will be monitored electronically, but no intervention will be applied. This will give participants time to become familiar with the e-pillbox and provide pre-intervention adherence data. All participants will receive a text message from study staff 1 week after initiation of the run-in to check-in on how they are doing with the e-pillbox. If a participant is experiencing difficulties, staff will offer assistance by phone. The first intervention will occur at 4 weeks (+/- 1 wk.). At this visit, participants will meet via video conferencing (or in person, if possible) with the coach. Participants at adherence intervention sites will begin the adherence-promoting intervention, including activation of dose reminders from the e-pillbox (as desired) and access to the adherence-tracking website. Participants at healthy living education intervention sites will begin the healthy living intervention, but will have no dose reminders from the e-pillbox and will not have access to the adherence-tracking website. The healthcare team will provide the usual level of care to all participants. Participants will have virtual (or phone) contact with coaches at increasing intervals between initiation of the intervention at week 4 and exit at week 14. The first check-in will occur at week 6 (+/- 1 wk), 2 weeks after initiation of the adherence-promoting intervention, the second will occur at week 10 (+/- 1 wk). This will allow intervals of increasing frequency between contacts as participants become more comfortable with procedures.

Parent participants: Parents of patient participants under 18 will be invited to participate in the study and accompany their child to study visits. Participating parents will be present at the beginning of the baseline visit to help their child provide demographic information. The parent will return at the end of the baseline visit, to learn how to use the e-pillbox (along with their child), to watch the educational videos and to respond to the PMBS and C-ATR. Parent participants will respond to the PMBS and C-ATR once more at week 14. Participating parents at adherence intervention sites will be present in the formation of the patient's action plan and choose their own action plan to support their child's adherence or independence. Parental participation throughout the study is encouraged but not mandatory.

HCP Participants: HCP-participants at adherence intervention sites will be trained to use the adherence-tracking website within 2 weeks before to 1 week after the first patient at their site completes the 4-week visit. HCP participants will be given access to the adherence data of all patient participants at their coaching site and invited to consult the website as often as they wish. HCP participants will also be shown a short (5 min) video providing education on assessing and supporting adherence.

HCP participants at adherence intervention sites will be advised that they will be informed by study staff about adherence events among participants in the interval between 4 and 14 weeks. When coaches review each participant's adherence on the portal during study visits, they will discuss non-adherence events with patients to determine if these were related to technical issues or real adherence issues. Within 1 week of study visits, the coach will provide the HCP with a copy of the patient's adherence calendar with a note as to whether the events seem to reflect real non-adherence. HCP will be advised that they will be under no obligation to act on this information, but may if they wish; if the participating HCP receiving information about a patient is not that patient's primary transplant care provider, they will be asked to transmit the information to the appropriate HCP on the patient's care team. Study staff will be provided with a suggested algorithm to follow if they receive such an alert.Within 2 weeks after the last patient at the site completes the 14-week visit at adherence intervention sites, HCP participants will complete questionnaires on their experience using the adherence-tracking web portal.

ELIGIBILITY:
Patient Inclusion Criteria

* kidney-only transplant recipients, who are ≥3 months post-transplant
* Aged 12 to 24 years
* Patients followed at one of the study sites

Patient Exclusion Criteria

* Patients with significant neurocognitive disabilities limiting their ability to understand and participate in their own care (as judged by the parents and the healthcare team)
* Patients unable to communicate in English or French (Montreal sites only)
* Multi-organ transplant recipients
* Patient has a sibling participating in Stage 3
* Patients with no internet access

Parents Inclusion Criteria • Parent of prevalent kidney-only transplant recipients 12-17 y (followed in a participating transplant center) will be eligible

Parents Exclusion Criteria

• Parents of patients 18-24 years old will be excluded as the older aged group is expected to be primarily responsible for their own care, independent of their parents. One parent per family will be eligible to avoid redundant representation.

Health Care Professionals Inclusion Criteria

* Representatives from the variety of disciplines typically involved in promoting medication adherence as deemed appropriate from each center.
* HCP from adherence intervention sites

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Taking Adherence | 14 weeks
  percentage of prescribed doses taken each day (as measured by electronic monitoring). The daily taking adherence score could take a value of 0%, 50%, or 100% for patients on twice-daily dosing, and 0% or 100% for patients on once-daily dosing. Each patient will have a taking adherence score for every day of observation (repeated measures). On days that the pillbox was not in use due to technical problems or participant non-use, no score will be given. To summarize adherence for each arm, the total percentage of days of observation for which there was 100% taking adherence will be calculated. The denominator for this calculation will be the total number of days of observation of each participant summed across all participants; the numerator will be the total number of days of observation of each participant for which taking adherence was 100% summed across all participants.
Timing Adherence | 14 weeks
  percentage of doses taken within 2 hours before to 2 hours after the prescribed dosing time each day (as measured by electronic monitoring). The daily timing adherence score could take a value of 0%, 50%, or 100% for patients on twice-daily dosing, and 0% or 100% for patients on once-daily dosing. Each patient will have a timing adherence score for every day of observation (repeated measures). On days that the pillbox was not in use due to technical problems or participant non-use, no score will be given. To summarize timing adherence for each arm, the total percentage of days of observation for which there is 100% timing adherence will be calculated. The denominator for this calculation will be the total number of days of observation of each participant summed across all participants; the numerator will be the total number of days of observation of each participant for which timing adherence is 100% summed across all participants.

SECONDARY OUTCOMES:
Self-reported Taking Adherence | 14 weeks (at baseline, 4-week, 6-week, 10-weeks, 14-week visits)
  Self-reported taking adherence will be assessed using the Basel Assessment of Adherence to Immunosuppressive Medications (BAASIS). Participants who report any missed doses in the prior 4 weeks will be classified as non-adherent; those missing no doses will be classified as adherent. Participants will also report the proportion of prescribed doses taken in the past 4 weeks (0-100%); a higher proportion indicates better taking adherence.
Self-reported Timing Adherence | 14 weeks (at baseline, 4-week, 6-week, 10-weeks, 14-week visits)
  Self-reported timing adherence will be assessed using the Basel Assessment of Adherence to Immunosuppressive Medications (BAASIS). Participants who report any late or missed doses in the prior 4 weeks will be classified as non-adherent; those with no late or missing doses will be classified as adherent. Participants will also report the proportion of prescribed doses taken on schedule in the past 4 weeks (0-100%); a higher proportion indicates better taking adherence.

OTHER OUTCOMES:
Recruitment feasibility: number of participants enrolled at each site | 3 months
  number of participants enrolled at each site
Acceptability of e-pillbox: PSSUQ | 14 weeks
  Ratings of participants on the Post-Study System Usability questionnaires (PSSUQ). The minimum score is 1 and the maximum 7. A lower score indicates better acceptability.
Acceptability of tracking website: PSSUQ | 10 weeks
  Ratings of participants on the Post-Study System Usability questionnaires (PSSUQ). The minimum score is 1 and the maximum 7. A lower score indicates better acceptability.
Drop out rate | 14 weeks
  proportion of participants who do not complete the 14-week study
Frequency that healthcare professionals access the tracking website | 10 weeks
  number of website accesses per patient per month
Frequency that patients/parents access the tracking website | 10 weeks
  number of website accesses per patient per month
Total time spent with the coach | 14 weeks
  total number of contact minutes (text, phone and in-person) with the study coach

CONTACTS AND LOCATIONS:
Overall Officials: Bethany J Foster, MD, MSCE, Principal Investigator — Montreal Children's Hospital of the MUHC; Annette DeVito Dabbs, PhD, Principal Investigator — University of Pittsburgh Medical Center
Locations (8):
- United States (4):
  - St-Louis Children's Hospital, St Louis, Missouri
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington
- Canada (4):
  - BC Children's Hospital, Vancouver, British Columbia
  - University of Toronto Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - CHU Ste-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Data generated will be available for use to other investigators in the research community. Data may be used for hypothesis testing, and to generate preliminary data in support of future research projects. A Data Sharing Committee, composed site investigators will review requests submitted for use of the data. If the request is approved, the appropriate data analysis will be performed and the results sent to the requesting investigator. Alternatively, depending on the request, it may be more appropriate to provide the requesting investigator with certain segments of the data. If this is the case, a file of the requested data (de-identified) will be provided to the investigator
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 12 months of publication of the study's main findings.
Access Criteria: Request for data submitted in writing. May require payment for costs associated with extracting the required data.